CLINICAL TRIAL: NCT01870739
Title: A Randomized, Double-blind, Active-controlled, Parallel Group, 52-week Study to Evaluate the Effect of LCZ696 Compared to Olmesartan on Regional Aortic Stiffness in Subjects With Essential Hypertension
Brief Title: A Study to Evaluate the Effect of LCZ696 on Aortic Stiffness in Subjects With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696A2224; 2012-005720-15 (EudraCT Number)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
Keywords: LCZ696,; Hypertension,; Aortic stiffness,; Central blood pressure,; Cardiovascular MRI
MeSH Terms: conditions — Hypertension | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; olmesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sacubitril/valsartan (LCZ696) (Experimental): Single drug treatment period: Patients received LCZ696 200mg once daily (q.d.) + placebo to 20 mg olmesartan q.d for 2 weeks. After 2 weeks, patients were dosed at the maintenance dose level (400 mg qd LCZ696 + placebo to 40 mg qd olmesartan) for 10 weeks.
  Add-on Period: After 12 weeks on single-drug treatment, patients continued in the study on the blinded maintenance dose and if required, open label amlodipine (2.5 mg, 5 mg, or 10 mg qd) was added to the treatment regimen and titrated according to the investigator's discretion to achieve target blood pressure.
  Interventions: Drug: sacubitril/valsartan (LCZ696); Other: placebo to olmesartan; Drug: Amlodipine (Optional)
- olmesartan (Active Comparator): Single drug treatment period: Patients received 20 mg olmesartan q.d + placebo to LCZ696 200mg once daily (q.d.) for 2 weeks. After 2 weeks, patients were dosed at the maintenance dose level (40 mg olmesartan q.d + placebo to 400 mg qd LCZ696) for 10 weeks.
  Add-on Period: After 12 weeks on single-drug treatment, patients continued in the study on the blinded maintenance dose and if required, open label amlodipine (2.5 mg, 5 mg, or 10 mg qd) was added to the treatment regimen and titrated according to the investigator's discretion to achieve target blood pressure.
  Interventions: Drug: olmesartan; Other: placebo to sacubitril/valsartan (LCZ696); Drug: Amlodipine (Optional)

INTERVENTIONS:
Drug: sacubitril/valsartan (LCZ696) — 200 mg tablets
  Arms: sacubitril/valsartan (LCZ696)
Drug: olmesartan
  Arms: olmesartan
Other: placebo to sacubitril/valsartan (LCZ696) — placebo
  Arms: olmesartan
Other: placebo to olmesartan — placebo
  Arms: sacubitril/valsartan (LCZ696)
Drug: Amlodipine (Optional) — If required, open label amlodipine (2.5 mg, 5 mg, or 10 mg qd) was added to treatment regimen

SUMMARY:
This was the first evaluation of the effects of LCZ696 on local and regional measures of aortic stiffness in subjects with mild to moderate hypertension and widened pulse pressure. The results of this exploratory study will help to understand the mechanism of action of LCZ696 and used to inform the design of future clinical studies with LCZ696 in subjects with cardiovascular diseases.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with essential hypertension, untreated or currently taking antihypertensive therapy

Key exclusion Criteria:

* women of child bearing potential (WOCBP) if not on highly effective contraception
* Malignant or severe hypertension (grade 3 of WHO classification)
* History or evidence of a secondary form of hypertension
* Transient ischemic cerebral attack (TIA) during the 12 months prior to screening or any history of stroke.
* Previous or current diagnosis of heart failure (New York Heart Association Class II-IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
- Novartis Investigative Site, Basel, Switzerland
- Novartis Investigative Site, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Hrabak-Paar M, Kircher A, Al Sayari S, Kopp S, Santini F, Schmieder RE, Kachenoura N, Yates D, Langenickel T, Bremerich J, Heye T. Variability of MRI Aortic Stiffness Measurements in a Multicenter Clinical Trial Setting: Intraobserver, Interobserver, and Intracenter Variability of Pulse Wave Velocity and Aortic Strain Measurement. Radiol Cardiothorac Imaging. 2020 Apr 30;2(2):e190090. doi: 10.1148/ryct.2020190090. eCollection 2020 Apr. PMID 33778551
- [Derived] Santini F, Pansini M, Hrabak-Paar M, Yates D, Langenickel TH, Bremerich J, Bieri O, Schubert T. On the optimal temporal resolution for phase contrast cardiovascular magnetic resonance imaging: establishment of baseline values. J Cardiovasc Magn Reson. 2020 Oct 5;22(1):72. doi: 10.1186/s12968-020-00669-1. PMID 33012283
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=32

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 115 patients were enrolled. One patient was discontinued after randomization before receiving any dose of study randomized medication.
  A total of 114 patients received study randomized medication
Groups:
- Sacubitril/Valsartan (LCZ696): LCZ696 based treatment strategy (LCZ696 200 mg for 2 weeks as initiation dose, LCZ696 400 mg for additional 50 weeks as maintenance dose. Optional amlodipine 2.5 to 10 mg add-on after Week 12 to reach blood pressure target)
- Olmesartan: Olmesartan based treatment strategy (olmesartan 20 mg for 2 weeks as initiation dose, olmesartan 40 mg for additional 50 weeks as maintenance dose. Optional amlodipine 2.5 to 10 mg add-on after Week 12 to reach blood pressure target)
Period: Single Drug Treatment (12 Weeks)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Started | 57 ("Start" = Safety/Pharmacokinetic/Pharmacodynamic analysis set) | 57
Initiation Dose Completed | 57 | 56
Maintenance Dose Started | 57 | 56
Completed | 54 ("Completed" indicates maintenance dose complete) | 53
Not Completed | 3 | 4
Not completed — Protocol deviation | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Administrative problems | 3 | 2
Period: Add-on Period (40 Weeks)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Started | 54 | 53
Completed | 51 | 51
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0
Not completed — Protocol deviation | 1 | 1
Not completed — Patient withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All patients that received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (7.8) | 59.2 (13.1) | 59.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ascending Aorta Distensibility at 52 Week
Description: Cardiovascular magnetic resonance imaging (MRI) scans were obtained at baseline prior to randomization, at week 52 for the assessment of local aortic distensibility. Ascending aorta distensibility was one of the 3 components for measuring local arota distensibility.
Time Frame: Baseline, 52 weeks
Population: Pharmacodynamic (PD) analysis set: All patients with any available PD data, who received any study drug and experienced no protocol deviations with relevant impact on PD data. Patients with both baseline and week 52 data were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: 10^(-3) x mmHg^(-1)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 49 | 53
10^(-3) x mmHg^(-1) | 0.269 (0.1283) | 0.330 (0.1233)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Olmesartan; Test type: Superiority or Other; p = 0.7324, Linear Model; Treatment as fixed effect and corresponding baseline as covariate; Mean Difference (Net) = -0.0616, 95% CI 2-sided [-0.4178 to 0.2947]

2. Primary Outcome: Change From Baseline in Proximal Descending Aorta Distensibility at 52 Weeks
Description: Cardiovascular magnetic resonance imaging (MRI) scans were obtained at baseline prior to randomization, at week 52 for the assessment of local aortic distensibility. Proximal descending aorta distensibility was one of the 3 components for measuring local arota distensibility.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 10^(-3) x mmHg^(-1)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 49 | 53
10^(-3) x mmHg^(-1) | 0.510 (0.1528) | 0.547 (0.1469)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Olmesartan; Test type: Superiority or Other; p = 0.8614, Linear Model; Treatment as a fixed effect and corresponding baseline as a covariate; Mean Difference (Net) = -0.0371, 95% CI 2-sided [-0.4582 to 0.3839]

3. Primary Outcome: Change From Baseline in Distal Descending Aorta Distensibility at 52 Weeks
Description: Cardiovascular magnetic resonance imaging (MRI) scans were obtained at baseline prior to randomization, at week 52 for the assessment of local aortic distensibility. Distal descending aorta distensibility was one of the 3 components for measuring local arota distensibility.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 10^(-3) x mmHg^(-1)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 49 | 53
10^(-3) x mmHg^(-1) | 0.417 (0.2242) | 0.498 (0.2156)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Olmesartan; Test type: Superiority or Other; p = 0.7946, Linear Model; Treatment as a fixed effect and corresponding baseline as a covariate; Mean Difference (Net) = -0.0812, 95% CI 2-sided [-0.6987 to 0.5362]

4. Secondary Outcome: Change From Baseline in Local Aortic Strain at 52 Weeks
Description: Cardiovascular magnetic resonance imaging (MRI) scans were obtained at baseline prior to randomization, at week 52 for the assessment of local aortic strain. Local aortic strain was measured by assessing ascending aorta strain, proximal descending aorta strain and distal descending aorta strain.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 49 | 53
percent
  Ascending Aorta Strain | -0.830 (0.7903) | 0.453 (0.7598)
  Proximal Descending Aorta Strain | -0.284 (0.8940) | -0.066 (0.8596)
  Distal Descending Aorta Strain | -1.092 (1.0956) | 0.225 (1.0533)

5. Secondary Outcome: Change From Baseline in Regional Aortic Pulse Wave Velocity at 52 Weeks
Description: Cardiovascular magnetic resonance imaging (MRI) scans were obtained at baseline prior to randomization, at week 52 for the assessment of regional aortic pulse wave velocity.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 49 | 53
meters per second (m/s) | -2.086 (0.5029) | -1.085 (0.4835)

6. Secondary Outcome: Change From Baseline in Central Blood Pressure at 52 Weeks
Description: Central blood pressure was determined by measuring central systolic blood pressure , diastolic blood pressure and pulse pressure.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 50 | 50
mmHg
  Central systolic blood pressure | -16.655 (1.4968) | -13.625 (1.4968)
  Central diastolic blood pressure | -10.318 (1.0578) | -10.432 (1.0578)
  Central pulse pressure | -6.539 (0.9428) | -3.041 (0.9428)

7. Secondary Outcome: Change From Baseline in Augmentation Pressure at 52 Weeks
Description: Augmentation pressure is the added pressure during systole due to wave reflection.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 50 | 50
mmHg | -2.443 (0.5950) | -1.437 (0.5950)

8. Secondary Outcome: Change From Baseline in Augmentation Index at 52 Weeks
Description: Augmentation index (Alx) is the percentage of the central pulse pressure due to wave reflection.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 50 | 50
percent | -2.385 (1.1805) | -1.515 (1.1805)

9. Secondary Outcome: Change From Baseline in Carotid-femoral Pulse Wave Velocity at 52 Weeks
Description: For pulse wave velocity calculation, the pressure waveform at the femoral site (using a partially inflated custom blood pressure cuff) and the carotid site (using hand -held applanation tonometry) were measured simultaneously. Pulse wave analysis was performed on the central aortic pressure waveform as derived from the brachial pressure waveform recorded in a partially-inflated blood pressure cuff around the upper arm.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Sacubitril/Valsartan (LCZ696) | Olmesartan
Number analyzed (Participants) | 50 | 50
meters per second (m/s) | -0.428 (0.1663) | -0.434 (0.1663)

10. Secondary Outcome: Number of Patients With Reported Adverse Events, Serious Adverse Events and Death
Description: This outcome measure summarizes patients with any adverse events, serious adverse events and death.
Time Frame: 12 weeks
Population: Safety analysis set: All patients that received study drug
Measure: Number; unit: Patients
Groups:
- Initiation Dose : Sacubitril/Valsartan (LCZ696 200mg): Patients received LCZ696 200 mg for 2 weeks as initiation dose for 2 weeks
- Initiation Dose: Olmesartan 20mg: Patients received olmesartan 20 mg for 2 weeks as initiation dose for 2 weeks
- Maintenance Dose: Sacubitril/Valsartan (LCZ696 400mg): After 2 weeks on initiation dose, patients were dosed at the maintenance dose level of LCZ696 400 mg for 10 weeks
- Maintenance Dose: Olmesartan 40 mg: After 2 weeks on initiation dose, patients were dosed at the maintenance dose level of olmesartan 40 mg for 10 weeks
- Sacubitril/Valsartan (LCZ696 400mg) +/- Amlodipine; Olmesartan 40mg +/- Amlodipine: Optional amlodipine 2.5 to 10 mg add-on after Week 12 to reach blood pressure target
Arm/Group | Initiation Dose : Sacubitril/Valsartan (LCZ696 200mg) | Initiation Dose: Olmesartan 20mg | Maintenance Dose: Sacubitril/Valsartan (LCZ696 400mg) | Maintenance Dose: Olmesartan 40 mg | Sacubitril/Valsartan (LCZ696 400mg) +/- Amlodipine | Olmesartan 40mg +/- Amlodipine
Number analyzed (Participants) | 57 | 57 | 57 | 56 | 54 | 53
Patients
  Any Adverse events | 13 | 16 | 21 | 28 | 31 | 38
  Serious Adverse Events | 0 | 2 | 0 | 2 | 6 | 5
  Death | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Initiation Dose : Sacubitril/Valsartan (LCZ696 200mg) | Initiation Dose: Olmesartan 20mg | Maintenance Dose: Sacubitril/Valsartan (LCZ696 400mg) | Maintenance Dose: Olmesartan 40 mg | Sacubitril/Valsartan (LCZ696 400mg) +/- Amlodipine | Olmesartan 40mg +/- Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/57 | 2/57 | 0/57 | 2/56 | 6/54 | 5/53
Other Adverse Events (participants affected / at risk) | 3/57 | 6/57 | 10/57 | 14/56 | 16/54 | 24/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initiation Dose : Sacubitril/Valsartan (LCZ696 200mg) (N=57) | Initiation Dose: Olmesartan 20mg (N=57) | Maintenance Dose: Sacubitril/Valsartan (LCZ696 400mg) (N=57) | Maintenance Dose: Olmesartan 40 mg (N=56) | Sacubitril/Valsartan (LCZ696 400mg) +/- Amlodipine (N=54) | Olmesartan 40mg +/- Amlodipine (N=53)
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fat necrosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initiation Dose : Sacubitril/Valsartan (LCZ696 200mg) (N=57) | Initiation Dose: Olmesartan 20mg (N=57) | Maintenance Dose: Sacubitril/Valsartan (LCZ696 400mg) (N=57) | Maintenance Dose: Olmesartan 40 mg (N=56) | Sacubitril/Valsartan (LCZ696 400mg) +/- Amlodipine (N=54) | Olmesartan 40mg +/- Amlodipine (N=53)
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2 | 4 | 5 | 11 | 10
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5 | 1 | 5
Dizziness (Nervous system disorders) | 1 | 2 | 4 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 6 | 2 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.